CLINICAL TRIAL: NCT01945242
Title: Nesina Tablets Special Drug Use Surveillance "Type 2 Diabetes Mellitus: Combination Therapy With Thiazolidinediones"
Brief Title: Alogliptin Tablets Special Drug Use Surveillance "Type 2 Diabetes Mellitus: Combination Therapy With Thiazolidinediones"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 121-012; JapicCTI-132265 (Registry Identifier: JapicCTI); JapicCTI-R150770 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes Melitus
Keywords: Drug Therapy
MeSH Terms: interventions — alogliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alogilptin 25mg, tablets, orally, once daily, up to 12 months
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: Nesina; SYR-322

SUMMARY:
The purpose of this study is to determine the safety and efficacy of long-term combination therapy with alogliptin (Nesina) and thiazolidinediones in patients with type 2 diabetes mellitus who failed to respond adequately to treatment with thiazolidinediones in addition to diet therapy and exercise therapy.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of alogliptin with a 1-year (12-month) observational period, designed to investigate the safety and efficacy of long-term combination therapy with alogliptin and thiazolidinediones in patients with type 2 diabetes mellitus in a routine clinical setting.

Participants will be patients with type 2 diabetes mellitus who failed to respond adequately to treatment with thiazolidinediones in addition to diet therapy and exercise therapy. The planned sample size is 1,000 subjects.

The usual adult dosage for oral use is 1 alogliptin tablet (25 mg) once daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not adequately respond to the following treatment • Treatment with thiazolidinediones in addition to diet therapy and exercise therapy

Exclusion Criteria:

* Patients contraindicated for Nesina

  1. Patients with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus (these patients require prompt adjustment of hyperglycemia by fluid infusion and insulin, and hence use of Nesina is not appropriate.)
  2. Patients with severe infection, pre- or post-operative patients, or patients with serious traumatic injury (blood glucose control by insulin injection is desirable for these patients, and hence use of Nesina is not appropriate.)
  3. Patients with a history of hypersensitivity to any ingredient of Nesina

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus who have been examined at a medical institution
Sampling Method: Non-Probability Sample
Enrollment: 1374 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 252 investigative site in Japan from 25 March 2011 to 30 June 2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus who failed to respond adequately to treatment receiving thiazolidinediones were enrolled in 1 of 2 treatment groups as follows: alogliptin + thiazolidinediones; alogliptin + other.
Groups:
- Alogliptin + Thiazolidinedione: Alogliptin 25 milligram (mg), tablets, orally, once daily for up to 12 months in participants who received a thiazolidinedione within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin.
- Alogliptin + Other: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months in participants who did not receive a thiazolidinedione within 3 months from the start of administration of alogliptin or during the treatment period of alogliptin.
Period: Overall Study
Arm/Group | Alogliptin + Thiazolidinedione | Alogliptin + Other
Started | 1251 | 123
Completed | 1248 | 120
Not Completed | 3 | 3
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin + Thiazolidinedione | Alogliptin + Other | Total
Number analyzed (Participants) | 1248 | 120 | 1368
Age, Customized [Number; unit: participants]
  Less than (<) 20 years | 1 | 0 | 1
  20-29 years | 5 | 0 | 5
  30-39 years | 29 | 4 | 33
  40-49 years | 120 | 12 | 132
  50-59 years | 214 | 22 | 236
  60-69 years | 412 | 35 | 447
  70-79 years | 337 | 39 | 376
  Greater than equal to (>=) 80 years | 130 | 8 | 138
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 462 | 41 | 503
  Male | 786 | 79 | 865
Body Mass Index [Number; unit: participants]
  <18.5 kilogram/square meter (kg/m^2) | 16 | 0 | 16
  >=18.5 to <25 kg/m^2 | 318 | 26 | 344
  >=25 to <30 kg/m^2 | 353 | 31 | 384
  >=30 kg/m^2 | 134 | 16 | 150
  Unknown | 427 | 47 | 474
Waist Circumference [Number; unit: participants]
  <85 centimeter (cm) (Male) | 60 | 7 | 67
  >=85 cm (Male) | 184 | 17 | 201
  Unknown (Male) | 542 | 55 | 597
  <90 cm (Female) | 92 | 4 | 96
  >=90 cm (Female) | 49 | 4 | 53
  Unknown (Female) | 321 | 33 | 354
Pregnancy Status [Number; unit: participants] — The baseline characteristic was analyzed only in female participants.
  participants
    Not pregnant | 462 | 41 | 503
    Pregnant | 0 | 0 | 0
Healthcare category [Number; unit: participants] — Participants were categorized as outpatient, inpatient, and outpatient and Inpatient (participants who were both outpatient and inpatient at any time prior to enrollment).
  participants
    Outpatient | 1209 | 120 | 1329
    Inpatient | 11 | 0 | 11
    Outpatient and Inpatient | 28 | 0 | 28
Health-related Complications [Number; unit: participants] — Participants were asssed on the basis of primary illness (had complications and had no complications) at the start of study.
  participants
    Had Complications | 1064 | 96 | 1160
    Had No Complications | 184 | 24 | 208
Diabetic complications [Number; unit: participants]
  Had Diabetic Complications | 203 | 15 | 218
  Had No Diabetic Complications | 1045 | 105 | 1150
Breakdown of diabetic complications [Number; unit: participants] — The baseline characteristic was analyzed only in participants who had diabetic complications. Participants could be counted in more than 1 category (including duplicates).
  participants
    Diabetic nephropathy | 128 | 5 | 133
    Diabetic retinopathy | 65 | 9 | 74
    Diabetic neuropathy | 71 | 6 | 77
Complications of Hypertension [Number; unit: participants]
  Had Hypertension Complications | 760 | 69 | 829
  Had No Hypertension Complications | 488 | 51 | 539
Complications of Dyslipidemia [Number; unit: participants]
  Had Dyslipidemia Complications | 766 | 63 | 829
  Had No Dyslipidemia Complications | 482 | 57 | 539
Complications of Hyperuricemia [Number; unit: participants]
  Had Hyperuricemia Complications | 106 | 10 | 116
  Had No Hyperuricemia Complications | 1142 | 110 | 1252
Complications of Liver Damage [Number; unit: participants]
  Had Liver Damage Complications | 200 | 18 | 218
  Had No Liver Damage Complications | 1048 | 102 | 1150
Breakdown of Complications of Liver Damage [Number; unit: participants] — Liver damage complications were categorized as hepatic steatosis, hepatitis alcoholic, chronic hepatitis, hepatic cirrhosis and any other complications related to liver damage. The baseline characteristic was analyzed only in participants who had liver damage complications. Participants could be counted in more than 1 category (including duplicates).
  participants
    Hepatic steatosis | 158 | 14 | 172
    Hepatitis alcoholic | 18 | 1 | 19
    Chronic hepatitis | 17 | 2 | 19
    Hepatic cirrhosis | 5 | 0 | 5
    Other | 8 | 2 | 10
Degree of Hepatic Dysfunction [Number; unit: participants] — Severity was determined using aspartate aminotransferase (AST) or alanine transaminase (ALT) values at the start of treatment with alogliptin. For the assessment of severity, the following categories were used and higher grades of serum AST or ALT were adopted.
  Normal: <50 international units per liter (IU/L) Grade 1: >=50 to <100 IU/L Grade 2: >=100 to <500 IU/L Grade 3: >=500 IU/L
  participants
    Normal | 769 | 74 | 843
    Grade 1 | 89 | 10 | 99
    Grade 2 | 11 | 0 | 11
    Grade 3 | 0 | 0 | 0
    Unknown | 379 | 36 | 415
Complications of Renal Damage [Number; unit: participants]
  Had Renal Damage Complications | 138 | 5 | 143
  Had No Renal Damage Complications | 1110 | 115 | 1225
Breakdown of Complications of Renal Damage [Number; unit: participants] — Renal damage complications were categorized as nephrotic syndrome, glomerulonephritis,renal failure chronic and any other complications related to renal damage. The baseline characteristic was analyzed only in participants who had renal damage complications. Participants could be counted in more than 1 category (including duplicates).
  participants
    Nephrotic syndrome | 1 | 0 | 1
    Glomerulonephritis | 3 | 0 | 3
    Renal failure chronic | 8 | 0 | 8
    Other | 126 | 5 | 131
Degree of Renal Dysfunction [Number; unit: participants] — Estimated glomerular filtration rate (eGFR) was calculated using variables of gender, age at the start of treatment, and serum creatinine values, and severity was determined based on the following categories. If the serum creatinine value at the start of treatment was not listed, the severity was reported as "unknown."
  Normal: >=90 milliliter per min (mL/min)/1.73^2 Mild: >=60 mL/min/1.73^2 to <90 mL/min/1.73^2 Moderate: >=30 mL/min/1.73^2 to <60 mL/min/1.73^2 Severe: <30 mL/min/1.73^2
  eGFR = 194 * Cr^-1.094 * (age)^-0.287 (* 0.739 if female) where Cr is creatinine clearance.
  participants
    Normal | 198 | 26 | 224
    Mild | 488 | 46 | 534
    Moderate | 174 | 15 | 189
    Severe | 10 | 0 | 10
    Unknown | 378 | 33 | 411
Complications of Heart Disease [Number; unit: participants]
  Had Heart Disease Complications | 142 | 9 | 151
  Had No Heart Disease Complications | 1106 | 111 | 1217
Breakdown of Complications of Heart Disease [Number; unit: participants] — Heart disease complications were categorized as Cardiac failure, Myocardial infarction, Angina pectoris, and any other complications related to heart disease. The baseline characteristic was analyzed only in participants who had heart disease complications. Participants could be counted in more than 1 category (including duplicates).
  participants
    Cardiac failure | 16 | 2 | 18
    Myocardial infarction | 27 | 3 | 30
    Angina pectoris | 71 | 4 | 75
    Other | 42 | 3 | 45
Complications of Heart Failure [Number; unit: participants]
  Had Heart Failure Complications | 16 | 2 | 18
  Had No Heart Failure Complications | 1232 | 118 | 1350
New York Heart Association (NYHA) Heart Failure Classification [Number; unit: participants] — NYHA functional classification ranges from Class I (participants with cardiac disease but without resulting limitations of physical activity), Class II (participants with cardiac disease resulting in slight limitation of physical activity), Class III (participants with cardiac disease resulting in marked limitation of physical activity), Class IV (participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). The baseline measure was analyzed only for participants who had complications of heart failure.
  participants
    NYHA Class I | 15 | 1 | 16
    NYHA Class II | 1 | 1 | 2
    NYHA Class III | 0 | 0 | 0
    NYHA Class IV | 0 | 0 | 0
Complications of Stroke-related Disease [Number; unit: participants]
  Had Stroke-related Disease Complication | 81 | 7 | 88
  Had No Stroke-related Disease Complication | 1167 | 113 | 1280
Breakdown of complications of stroke-related disease [Number; unit: participants] — The baseline characteristic was analyzed only in participants who had stroke-related disease complications. Participants could be counted in more than 1 category (including duplicates).
  participants
    Cerebral infarction | 80 | 7 | 87
    Transient ischemic attack | 1 | 0 | 1
Complications of Allergic Disease [Number; unit: participants]
  Had Allergic Disease Complication | 58 | 7 | 65
  Had No Allergic Disease Complication | 1190 | 113 | 1303
Breakdown of Complications of Allergic Disease [Number; unit: participants] — The baseline characteristic was analyzed only in participants who had allergic disease complications. Participants could be counted in more than 1 category (including duplicates).
  participants
    Asthma bronchial | 27 | 3 | 30
    Pollinosis | 12 | 0 | 12
    Rhinitis allergic | 25 | 4 | 29
    Dermatitis allergic | 2 | 0 | 2
Complications of Malignant Tumor [Number; unit: participants] — This baseline measure was analysed for participants who had malignant tumor at the start of the study.
  participants
    Had Malignant Tumor Complications | 13 | 5 | 18
    Had No Malignant Tumor Complications | 1235 | 115 | 1350
Complications of Malignant Tumor (narrow definition) [Number; unit: participants] — This baseline measure was analysed for participants who had malignant tumor and/or benign tumor at the start of the study.
  participants
    Had Malignant Tumor Complications | 11 | 2 | 13
    Had No Malignant Tumor Complications | 1237 | 118 | 1355
Other Complications [Number; unit: participants] — Participants who had complications other than diabetic, hypertension, dyslipidemia, hyperuricemia, liver damage, renal damage, heart disease, heart failure, stroke-related disease, allergic disease, and malignant tumor were analyzed.
  participants
    Had Other Complications | 376 | 34 | 410
    Had No Other Complications | 872 | 86 | 958
Presence of Medical History [Number; unit: participants] — The baseline characteristic was analysed in participants who had any illness (medical history of any previous illness) at the start of the study.
  participants
    Had Presence of Medical History | 162 | 19 | 181
    Had No Presence of Medical History | 960 | 88 | 1048
    Unknown | 126 | 13 | 139
History of Allergies [Number; unit: participants]
  Had History of Allergies | 78 | 7 | 85
  Had No History of Allergies | 1066 | 95 | 1161
  Unknown | 104 | 18 | 122
History of Alcohol Consumption [Number; unit: participants]
  Had Alcohol Consumption | 333 | 34 | 367
  Had No Alcohol Consumption | 690 | 60 | 750
  Unknown | 225 | 26 | 251
Smoking Classification [Number; unit: participants]
  Never Smoked | 525 | 45 | 570
  Current Smoker | 204 | 25 | 229
  Ex-smoker | 233 | 24 | 257
  Unknown | 286 | 26 | 312
Time from Diagnosis of Type 2 Diabetes [Number; unit: participants]
  <2 years | 158 | 35 | 193
  >=2 to <5 years | 187 | 17 | 204
  >=5 to <10 years | 247 | 21 | 268
  >=10 years | 288 | 22 | 310
  Unknown | 368 | 25 | 393
Glycosylated Hemoglobin A1c (HbA1c) [Number; unit: participants]
  HbA1c <6.0 percent | 30 | 3 | 33
  HbA1c >=6.0 to <7.0 percent | 289 | 27 | 316
  HbA1c >=7.0 to <8.0 percent | 461 | 44 | 505
  HbA1c >=8.0 percent | 365 | 36 | 401
  Unknown | 103 | 10 | 113

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. The safety analysis was planned to be assessed in alogliptin + thiazolidinedione and alogliptin + other arm separately.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Alogliptin + Thiazolidinedione | Alogliptin + Other
Number analyzed (Participants) | 1248 | 120
participants
  Hypothyroidism | 1 | 0
  Hyperglycaemia | 1 | 0
  Hypoglycaemia | 5 | 1
  Dyslipidaemia | 1 | 0
  Dizziness | 3 | 0
  Photopsia | 1 | 0
  Hypertension | 1 | 0
  Abdominal distension | 1 | 0
  Diarrhoea | 1 | 0
  Eczema | 1 | 0
  Pruritus | 1 | 0
  Arthralgia | 1 | 0
  Joint swelling | 1 | 0
  Local swelling | 1 | 0
  Pyrexia | 1 | 0
  Blood insulin decreased | 1 | 0
  Blood insulin increased | 1 | 0
  Hand fracture | 1 | 0
  Rib fracture | 1 | 0

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAEs) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The safety analysis was planned to be assessed in alogliptin + thiazolidinedione and alogliptin + other arm separately.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Alogliptin + Thiazolidinedione | Alogliptin + Other
Number analyzed (Participants) | 1248 | 120
participants
  Hyperglycaemia | 1 | 0
  Hypoglycaemia | 2 | 0

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of the thiazolidinedione treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to 12 months)
Population: The efficacy assessment population was defined as participants who completed the study and had available efficacy data at baseline and post baseline.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Alogliptin: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months.
Arm/Group | Alogliptin
Number analyzed (Participants) | 1129
percentage of glycosylated hemoglobin
  Baseline (n=1124) | 7.67 (1.179)
  Change at Month 1 (n=879) | -0.25 (0.597)
  Change at Month 3 (n=1005) | -0.47 (0.988)
  Change at Month 6 (n=988) | -0.53 (1.098)
  Change at Month 12 (n=949) | -0.64 (1.133)
  Change at Final assessment (n=1124) | -0.57 (1.143)

4. Secondary Outcome: Percentage of Participants of Achieving Objective Glycemic Control
Description: The rate of achieving objective glycemic control in HbA1c level, was calculated at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12). Glycemic control was measured as <8.0 percent, <7.0 percent, and <6.0 percent of glycosylated hemoglobin. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of the thiazolidinedione treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to 12 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin
Number analyzed (Participants) | 1129
percentage of participants
  <8.0 percent (Baseline) (n=1124) | 68.0 (1.179)
  <8.0 percent (Month 1) (n=879) | 75.8 (0.597)
  <8.0 percent (Month 3) (n=1005) | 84.2 (0.988)
  <8.0 percent (Month 6) (n=988) | 84.5 (1.098)
  <8.0 percent (Month 12) (n=949) | 87.1 (1.133)
  <8.0 percent (Final assessment) (n=1124) | 83.6 (1.143)
  <7.0 percent (Baseline) (n=1124) | 27.6
  <7.0 percent (Month 1) (n=879) | 34.3
  <7.0 percent (Month 3) (n=1005) | 47.1
  <7.0 percent (Month 6) (n=988) | 51.2
  <7.0 percent (Month 12) (n=949) | 57.5
  <7.0 percent (Final assessment) (n=1124) | 54.2
  <6.0 percent (Baseline) (n=1124) | 2.7
  <6.0 percent (Month 1) (n=879) | 3.2
  <6.0 percent (Month 3) (n=1005) | 5.6
  <6.0 percent (Month 6) (n=988) | 6.8
  <6.0 percent (Month 12) (n=949) | 8.2
  <6.0 percent (Final assessment) (n=1124) | 8.0

5. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change between the fasting blood glucose value collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of the thiazolidinedione treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to 12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Alogliptin
Number analyzed (Participants) | 1129
milligram per deciliter (mg/dL)
  Baseline (n=389) | 145.4 (41.25)
  Change at Month 1 (n=283) | -9.8 (35.39)
  Change at Month 3 (n=301) | -11.8 (37.63)
  Change at Month 6 (n=297) | -13.9 (41.75)
  Change at Month 12 (n=293) | -16.2 (35.46)
  Change at Final assessment (n=398) | -13.5 (40.25)

6. Secondary Outcome: Change From Baseline in Fasting Insulin
Description: The change between the fasting insulin value collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of the thiazolidinedione treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to 12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin
Number analyzed (Participants) | 1129
mg/dL
  Baseline (n=82) | 6.32 (3.121)
  Change at Month 1 (n=54) | 0.19 (1.519)
  Change at Month 3 (n=57) | -0.02 (1.946)
  Change at Month 6 (n=60) | 0.29 (3.505)
  Change at Month 12 (n=68) | -0.32 (1.980)
  Change at Final assessment (n=82) | -0.25 (1.951)

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin + Thiazolidinedione | Alogliptin + Other
Serious Adverse Events (participants affected / at risk) | 3/1248 | 0/120
Other Adverse Events (participants affected / at risk) | 11/1248 | 2/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + Thiazolidinedione (N=1248) | Alogliptin + Other (N=120)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + Thiazolidinedione (N=1248) | Alogliptin + Other (N=120)
Diabetes mellitus (Metabolism and nutrition disorders) | 11 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.